CLINICAL TRIAL: NCT03666520
Title: Inpatient Medications: Switching Medications From Intravenous to Oral
Brief Title: Switching Medications From Intravenous to Oral
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Robert Turer, Clinical Informatics Fellow, Vanderbilt University Medical Center
Other Study IDs: 023420
Record Dates: First submitted 2018-08-29; First posted 2018-09-11 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Physician's Role; Administration, Oral
Keywords: medication administration, IV to PO conversion; IV to PO conversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Clinician not prompted to change the drug from intravenous to oral equivalent.
- Cohort with clinician being prompted to convert drug: This arm would include the provider being prompted to change the intravenous drug to the oral equivalent.
  Interventions: Other: Clinical Decision Support prompted to the clinician to convert drug.

INTERVENTIONS:
Other: Clinical Decision Support prompted to the clinician to convert drug. — This study is designed to further research the conversion of Intravenous medications to oral medications in patients in an inpatient setting whenever it is appropriate and safe. We have chosen eight medications to research in this study. These medications were chosen because large difference in cost between an intravenous (IV) dose of this medication versus an oral (PO) dose of this medication exist. This study aims to further evaluate the appropriateness and safety of converting IV medications to PO medications for hospitalized patients through a pilot clinical trial.
  Groups: Cohort with clinician being prompted to convert drug

SUMMARY:
In a recent report, drug spending increased by 23.4 percent annually in the inpatient setting from 2013 to 2015 with the average inpatient drug spending increasing from $714 to $990 per admission. A retrospective analysis from Johns Hopkins showed potential annual savings of over $1,100,000 dollars with a switch from intravenous (IV) to oral (PO) administration of four inpatient medications. Another study actively encouraging the conversion of IV to PO medications demonstrated a decrease in therapeutic costs.

A number of benefits occur at the conversion of IV to oral medications including the reduced risk of secondary cannula- related infections, inflammation, and pain in the area of administration. Most oral agents are less expensive than the related IV medications. Other benefits occur in indirect administration costs such as the expense of nursing labor and equipment. The switch from IV to oral medication has also been shown to result in earlier discharge of patients, potentially saving medical costs.

The investigators have chosen to further the research of the conversion of IV to PO medications by combining prior knowledge on the subject with robust clinical decision support. Our research will prompt providers at the right time in the workflow to switch from IV to PO medications. The investigators will exclude patients less than 18 years old, with a NPO status, or a severe disease state (vasopressor dependent, decreased consciousness, seizures, severely immunocompromised (ANC < 500), or life- threatening infections such as sepsis, Central Nervous System (CNS) infections, endocarditis, osteomyelitis, etc.). The medications eligible for this research project were identified through comparison of the wholesale price of the intravenous and oral formulations. To select medications with a potential for savings, the investigators factored in the frequency of IV administrations in the past five months using our electronic health record system (EHR) to help identify highly utilized medications. The product of the largest cost differential and frequency was used to decide on the following list of medications for this project: Lacosamide, Doxycycline, Levothyroxine, Linezolid, Acetaminophen, Rifampin, Amiodarone and Levofloxacin.

The principal trigger for the clinical decision support prompt will be a current diet order listed in the patient's chart or an order for another medication via the oral route. These orders will flag the patient as eligible for po medications. Once the patient has been identified to be eligible for PO medications, the presence of an order for an IV formulation of one of the above drugs will prompt a once-daily alert to the provider upon opening the chart for the conversion to PO medication. Providers will be randomized to receive the alert. Past experience has shown that such an alert will remind providers not only to switch the drug in questions to PO form, but other medications as well. For the providers not receiving the alert, the investigators will record when it would have been triggered for the first time. The trial will run for three months to completion.

Analysis at the time of study completion will occur on primary (number of doses of candidate medication administered IV and PO after the alert) and secondary outcomes (number of doses of other medication not on our IV and PO list, cost savings, presence of an iv drip, episodes of sepsis or bacteremia). The investigators will monitor for potential complications by monitoring length of stay after triggering the alert. The investigators will also monitor the doses of hyaluronidase administered to patients after the alert was triggered.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient
* Over 18
* Able to tolerate oral medications
* Currently taking one of our eight medications under research intravenously

Exclusion Criteria:

* Children (<18)
* Unable to tolerate an oral medication (or NPO)
* Severe disease severity (Ex. vasopressor dependent, seizures, etc...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatient adult patients that are currently being given one of our 8 chosen drugs intravenously.
Sampling Method: Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Medication change from intravenous to oral | Change from Baseline to 4 months
  Number of doses of candidate medication administered intravenous and oral after the alert

SECONDARY OUTCOMES:
Doses of other medications | Change from Baseline to 4 months
  Number of doses of other medication not on our intravenous and oral list

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Lehmann, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided